CLINICAL TRIAL: NCT00087425
Title: A Phase II Trial Of Bryostatin-1 In Combination With Rituximab In Rituximab-Refractory Indolent B-cell Non Hodgkin's Lymphoma And Chronic Lymphocytic Leukemia
Brief Title: Bryostatin 1 and Rituximab in Treating Patients With B-Cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000377250; NIA-CII0301; NCI-6216
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2007-01

CONDITIONS: Leukemia; Lymphoma
Keywords: contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; recurrent grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; refractory chronic lymphocytic leukemia; Waldenström macroglobulinemia; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; bryostatin 1

INTERVENTIONS:
Biological: rituximab
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bryostatin 1, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Bryostatin 1 may help rituximab kill more cancer cells by making them more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving bryostatin 1 together with rituximab works in treating patients with B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia that has not responded to previous treatment with rituximab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and safety of bryostatin 1 and rituximab in patients with rituximab-refractory indolent B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia (CLL).
* Determine the antitumor response in patients treated with this regimen.

Secondary

* Determine the effects of this regimen on the functional and molecular status of effector cells (i.e., NK cells, monocytes, and dendritic cells) in these patients.
* Determine the expression of CD20 and complement-inhibitory molecules on tumor cells before and after treatment with this regimen in these patients.
* Determine the effects of this regimen on the global gene expression pattern in CLL cells of these patients.

OUTLINE: This is a multicenter study.

Patients receive bryostatin 1 IV continuously over 24 hours on days -6, 2, and 9 of course 1 and on days 2 and 9 of courses 2-6. Patients also receive rituximab IV over 4 hours on days 1, 8, 15, and 22 of courses 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 18-48 patients (9-24 with non-Hodgkin's lymphoma and 9-24 with chronic lymphocytic leukemia) will be accrued for this study within 12-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically or cytologically confirmed diseases:

  * Indolent B-cell non-Hodgkin's lymphoma (NHL)

    * Stage II-IV disease
  * Chronic lymphocytic leukemia (CLL) meeting 1 of the following risk criteria:

    * Intermediate-risk with progressive disease
    * High-risk, modified Rai stage disease
* CD20-positive by flow cytometry or immunohistochemistry
* Measurable disease
* Rituximab-refractory disease, defined as failure to achieve a response to the last course of prior treatment with rituximab alone or in combination with other therapeutic modalities
* No known neoplastic leptomeningeal involvement and/or brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 50,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal (unless due to Gilbert's disease or organ involvement by NHL or CLL)

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No history of anaphylaxis or immunoglobulin (Ig) E-mediated hypersensitivity to murine protein

  * Prior infusion reactions to rituximab without an IgE component allowed
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Radiotherapy
* At least 12 weeks since prior rituximab
* More than 4 weeks since prior immunotherapy and recovered

Chemotherapy

* No more than 3 prior chemotherapy regimens
* More than 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* No concurrent glucocorticoids

Radiotherapy

* At least 12 weeks since prior radioimmunotherapy
* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* At least 4 weeks since prior therapy for the malignancy
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Feasability and safety
Antitumor response

SECONDARY OUTCOMES:
Functional and molecular status of effector cells
Expression of CD20 and complement-inhibitory molecules on tumor cells before and after treatment
Effects on global gene expression pattern in chronic lymphocytic leukemia cells

CONTACTS AND LOCATIONS:
Overall Officials: Igor Espinoza-Delgado, MD, Study Chair — Gerontology Research Center
Locations (1):
- NIH - Warren Grant Magnuson Clinical Center, Bethesda, Maryland, United States